CLINICAL TRIAL: NCT02331823
Title: New Super-short Course Regimen for Retreatment Pulmonary Tuberculosis
Brief Title: Research on New Regimens for Retreatment Pulmonary Tuberculosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Shanghai Center for Disease Control and Prevention (Other); Jiangsu Province Centers for Disease Control and Prevention (Network); Zhejiang University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Qing Zhang, Chief physician, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013ZX10003009
Record Dates: First submitted 2014-12-31; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Reinfection Pulmonary Tuberculosis
MeSH Terms: interventions — Ethambutol; Pyrazinamide; Rifabutin; Moxifloxacin; Isoniazid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm A: super-short retreatment regimen (Experimental): A regimen of 5 drugs is to be administered. Isoniazid Aminosalicylate Tablets,0.3g tid po for 5 mon moxifloxacin tab, 0.4g qd po for 5 mon rifabutin capsule,0.3g qd po for 5 mon ethambutol tab, 0.75g qd po for 5 mon pyrazinamide tab, 0.5g tid po for 5 mon
  Interventions: Drug: Isoniazid Aminosalicylate Tablets
- arm B:standardized retreatment regimen (Active Comparator): 8-9 months of standardized regimen is to be administered. regimen 1.2SHREZ/6HRE streptomycin injectable,0.75g qd intramuscular for 2 mon isoniazid tab,0.3g qd po for 8 mon rifampicin capsule,0.45-0.6g po for 8 mon ethambutol tab, 0.75g qd po for 8 mon pyrazinamide tab, 0.5g tid po for 2 mon or regimen 2.3HREZ/6HRE isoniazid tab,0.3g qd po for 9 mon rifampicin capsule,0.45-0.6g po for 9 mon ethambutol tab, 0.75g qd po for 9 mon pyrazinamide tab, 0.5g tid po for 3 mon
  Interventions: Drug: Streptomycin injectable

INTERVENTIONS:
Drug: Isoniazid Aminosalicylate Tablets — a regimen consists of 5 anti-TB drugs (Isoniazid Aminosalicylate Tablets+pyrazinamide tablets+ethambutol tablets+rifabutin capsules+moxifloxacin tablets)to treat retreatment pulmonary tuberculosis patients. The total treatment course is 5 months.
  Other Names: ethambutol tablets; pyrazinamide tablets; rifabutin capsules; moxifloxacin tablets
  Arms: arm A: super-short retreatment regimen
Drug: Streptomycin injectable — standardized regimen 2 months of streptomycin injectable + isoniazid tablets + ethambutol tablets + rifampicin capsules + pyrazinamide tablets and 6 months of isoniazid tablets + ethambutol tablets + rifampicin capsules or 3 months of isoniazid tablets + ethambutol tablets + rifampicin capsules + pyrazinamide tablets and 6 months of isoniazid tablets + ethambutol tablets + rifampicin capsules to treat Arm B patients as a control to arm A.The treatment course is 8-9 months.
  Other Names: isoniazid tablets; ethambutol tablets; rifampicin capsules; pyrazinamide tablets
  Arms: arm B:standardized retreatment regimen

SUMMARY:
Multi-center, prospective study is performed to investigate the efficacy of new short-course regimen for retreatment pulmonary tuberculosis patients.

To obtain optimized short-course regimen, decrease treatment cost and improve success rate.

DETAILED DESCRIPTION:
China is the country with the second highest Tuberculosis (TB) burden in the world. Most of the retreatment TB patients may develop multi-drug resistant. The resistant rate of any of the anti-TB drug is 35.9%, and the multi-drug resistant rate is 15.4%. Retreatment TB becomes one of the factors which inhibit the decrease of morbidity and mortality of TB. It is also a tuff work in TB control. At present the standardized regimen for retreatment TB is 2SHREZ/6HRE or 3HREZ/6HRE. The drugs in the regimen are all first-line anti-TB drugs which are unsuitable for the high drug resistance prevalence, because the cure rate of this regimen is low and the adverse reaction is severe.

Our study is a national multi-center, prospective trail to investigate the efficacy of a new super-short regimen for retreatment TB patients. The new regimen consists of 5 drugs lasting 5 months. The cure rate and success rate of the new regimen is compared with standardized regimen usually 8-9 months in order to obtain the optimized regimen.

ELIGIBILITY:
Inclusion Criteria:

* Sputum confirmed diagnosis of retreatment pulmonary tuberculosis
* Must be able to swallow tablets
* Must be able to sign written informed consent form

Exclusion Criteria:

* Extra-pulmonary tuberculosis
* Diabetes
* Allergy to any of the medications in the regimen or pregnancy
* Liver disease
* Renal disease
* Metabolic disease
* Immune system disease
* Hematological disease
* Nervous system and mental disease
* Endocrine disease
* Malignant disease
* Receiving immunosuppressive therapy
* HIV/AIDS
* Alcohol addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
success rate | for arm A,the point is 5 month after treatment. For arm B,the time point is at the end of the 8 or 9 month's treatment.

SECONDARY OUTCOMES:
adverse reaction rate | for arm A,the point is 5 month after treatment. For arm B,the time point is at the end of the 8 or 9 month's treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Heping Xiao, M.D, Principal Investigator — Shanghai Pulmonary Hospital,China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yan L, Kan X, Zhu L, Xu K, Yin J, Jie L, Li Y, Yue J, Cui W, Du J, Wang L, Tan S, Jiang X, Zeng Z, Xu S, Wang L, Chen Y, He W, Gao X, Bai D, Zhao C, Yan X, Zhu Y, Fan Y, Xie L, Deng A, Zhang Q, Xiao H. Short-course Regimen for Subsequent Treatment of Pulmonary Tuberculosis: A Prospective, Randomized, Controlled Multicenter Clinical Trial in China. Clin Ther. 2018 Mar;40(3):440-449. doi: 10.1016/j.clinthera.2018.01.013. Epub 2018 Mar 6. PMID 29519716